CLINICAL TRIAL: NCT00921011
Title: Iron and Atherosclerosis: Longitudinal Study in Perimenopausal Women With Risk Factors for Atherosclerosis
Brief Title: Longitudinal Study in Perimenopausal Women With Risk Factors for Atherosclerosis
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Subha Raman, Professor of Medicine, Ohio State University
Other Study IDs: 2008H0308; R01HL095563 (NIH)
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Atherosclerosis
Keywords: hypertension; diabetes; smoking; hyperlipidemia; atherosclerosis risk
MeSH Terms: conditions — Atherosclerosis; Hypertension; Diabetes Mellitus; Smoking; Hyperlipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Perimenopausal women: Women at the beginning stages of menopause

SUMMARY:
The study hypothesis (or theory) is that monthly loss of iron before menopause may reduce women's risk of hardening of the arteries, or atherosclerosis.

This study uses noninvasive, noncontrast magnetic resonance imaging (MRI) of arteries in women entering menopause. This will help to determine if there is a correlation between iron accumulation and hardening of the arteries. In addition, blood levels of hormones will be measured to help show differences due to hormone levels vs. iron accumulation.

DETAILED DESCRIPTION:
Atherosclerosis, or hardening of the arteries, is the underlying disease responsible for the vast majority of cardiovascular morbidity and mortality and afflicted over 30 million Americans in 2005. While the prevalence of atherosclerosis is similar in women and men, women enjoy a ~5-10 year lag in onset of cardiovascular events compared to men. After menopause, a state defined by marked reduction in ovarian hormone production, the incidence of events such as heart attack and stroke caused by atherosclerotic plaque rises up to threefold regardless of age range. This has prompted numerous investigations of hormone therapy (HT) to lower cardiovascular risk to premenopausal levels. Therapeutic trials, however, have not realized a cardiovascular benefit; in fact, initiating HT in large randomized trials did not decrease and possibly increased cardiovascular risk. Studies of coronary heart disease prevention have shown mixed results using estrogen alone vs. estrogen plus progestin, while studies of stroke prevention have consistently shown increased risk with HT. Clearly, different therapeutic interventions warrant consideration. This proposal seeks to investigate a novel perspective using longitudinal clinical studies in women at risk of atherosclerosis. The studies involve a new noncontrast, noninvasive MRI method with blood tests that measure cholesterol, hormone levels, and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* women at least 40 yrs of age
* between 1 and 6 menstrual cycles in the past 12 months
* 2 or more of the following risk factors: high blood pressure, diabetes, high cholesterol, smoking
* no known heart or vascular disease

Exclusion Criteria:

* any known cardiovascular disease such as coronary disease, peripheral vascular disease, heart failure
* contraindication to MRI scan (e.g. aneurysm clip, iron-containing metal)

NOTE that orthopedic hardware is usually MRI-compatible. We will go over detailed screening before enrollment.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Perimenopausal women
Sampling Method: Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2009-05; Primary Completion 2018-02 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
vessel wall changes over time that precede plaque buildup | baseline, 1-year follow-up and 2-year follow-up

SECONDARY OUTCOMES:
development of cardiovascular disease | annually for 4 years after baseline visit

CONTACTS AND LOCATIONS:
Overall Officials: Subha V Raman, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State Univeristy Medical Center, Columbus, Ohio, United States